CLINICAL TRIAL: NCT05530317
Title: CArdiac REhabilitation for Building Exertional heArt Rate for Chronotropic Incompetence in Long COVID-19 (CARE BEAR-LC): A Proof-of-Concept, Mechanistic Trial
Brief Title: CArdiac REhabilitation for Building Exertional heArt Rate for Chronotropic Incompetence in Long COVID-19
Acronym: CARE BEAR-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37106
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Long COVID; COVID-19
Keywords: chronotropic incompetence; cardiac rehabilitation; cardiopulmonary exercise testing
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: pre- post-
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (Experimental): Participants will undergo 12 weeks of standard of care cardiac rehabilitation.
  Interventions: Behavioral: Cardiac Rehabilitation
- Control Arm (No Intervention): No intervention control group

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — Exercise prescriptions will be based on the heart rate performance during the baseline CPET. The intensity of the exercise prescription and level of monitoring will be tailored to the individual participant's performance on their baseline CPET according to guidelines. Exercise will be prescribed by a Cardiac Exercise Physiologist in accordance with standard cardiac rehabilitation protocols with special attention to post-exertional malaise. Resistance exercise activities will also be incorporated. Recumbent exercise will be utilized based on assessment by exercise physiologist and patient. Dietary counseling, smoking cessation counseling for smokers, and medication counseling will be incorporated according to standard cardiac rehabilitation protocols. Most participants will participate in a hybrid approach (12-16 sessions in person), but participants will be allowed to select a fully in-person approach (36 sessions).
  Arms: Cardiac Rehabilitation

SUMMARY:
The goal of this proof-of-concept clinical trial is to determine whether cardiac rehabilitation improves exercise capacity and chronotropic (heart rate) response to exercise among people with Long COVID. The study will include individuals with confirmed SARS-CoV-2 infection, symptoms not present prior to COVID-19 that are persistent for at least 3 months after acute infection ("Long COVID"), and who have reduced exercise capacity less than predicted and reduced heart rate response during cardiopulmonary exercise testing (CPET). In addition to the primary outcome of change in peak VO2, secondary outcomes will include change in symptoms including autonomic symptoms (COMPASS-31), anxiety (GAD-7), depression (PHQ-9), endothelial function with brachial artery flow-mediated dilation, and satisfaction (net-promotor score).

DETAILED DESCRIPTION:
Study Overview

This single-center, proof-of-concept mechanistic study of cardiac rehabilitation will use a pre-post design to establish whether there is any effect of cardiac rehabilitation on adjusted heart rate reserve achieved and peak oxygen consumption (peak VO2) in LC.

Once a participant is identified as potentially eligible, they will be contacted by the study team. Participants will be asked to co-enroll in the Long-term Impact of Infection with Novel Coronavirus observational cohort ("LIINC" NCT 04362150). If participants do not agree to be co-enrolled in LIINC (if they are not already included) and the Cardiovascular Sub-Study, they will not be allowed to enroll.

Participants will be consented by the PI or research team before any procedures take place. Participants who provide written informed consent and meet the inclusion criteria will be enrolled into the study. They undergo a series of baseline measurements as outlined in the Schedule of Events. They will participate in 12 weeks of cardiac rehabilitation and then undergo follow-up measurements to determine the safety, clinical impact, and biological impact of the therapy as outlined in the Schedule of Events.

Blood collection will occur at baseline and after completion of cardiac rehabilitation as per the Schedule of Events and will be timed to stay within Red Cross Guidelines (less than 480 mL every 8 weeks).

The details of the visit schedule are outlined below. Ultimately, the most up to date Schedule of Events will be the final guide for what events are to occur at each specific study visit.

Informed Consent

The study PI or their designee will explain the risks and benefits of the study and obtain written informed consent. Those who consent to participate in the study will undergo a Screening Assessment.

Screening Assessment

Assessments performed exclusively to determine eligibility for this study will be performed only after obtaining informed consent. Assessments performed for clinical indication (not exclusively to determine study eligibility) or other research studies may be used for screening even if the studies were performed before informed consent was obtained. For example, a screening cardiopulmonary exercise test may be used to establish eligibility that was performed through clinical practice or for research through the LIINC study or RECOVER. However, these measurements may be repeated at the discretion of the PI.

Following informed consent, study screening will occur during a period of one or more visits. The Screening Assessment will include a physical examination by a study clinician (physician, nurse, or physician assistant). Details of the participant's COVID-19 history will be reviewed and/or confirmed, and a symptom assessment will be performed.

Baseline Assessments

After consenting but prior to starting cardiac rehabilitation, all participants will undergo baseline assessments including symptom assessments, cardiopulmonary exercise testing and vascular function studies.

Intervention

Participants who screen into the study and complete baseline measurements will then start standard of care cardiac rehabilitation at University of California, San Francisco (UCSF) Parnassus Campus. Exercise prescriptions will be based on the heart rate performance during the baseline CPET. Standard clinical assessments will be made to tailor recommendations during the course of cardiac rehabilitation. The intensity of the exercise prescription and level of monitoring will be tailored to the individual participant's performance on their baseline CPET according to guidelines. Exercise will be prescribed by a Cardiac Exercise Physiologist in accordance with standard cardiac rehabilitation protocols. Resistance exercise activities will also be incorporated. Recumbent exercise will be utilized based on assessment by exercise physiologist and patient. Dietary counseling, smoking cessation counseling for smokers, and medication counseling will be incorporated according to standard cardiac rehabilitation protocols. Participants are asked to commit to attending at least 24 sessions, of which 12 (one per week for 12 weeks) must be in person at UCSF Parnassus. Participants will be allowed to select a fully in-person approach (36 sessions) or hybrid approach (12-24 in person, 12-24 virtual for up to 36 total sessions).

Duration of intervention: 12 weeks

Follow Up Assessments (Week 12) After completion of cardiac rehabilitation (approximately 12 weeks after start), participants will complete the follow up assessments within 2 weeks, which will include the same assessments as baseline as well as an assessment of satisfaction with cardiac rehabilitation as measured with the net-promotor score.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Previously documented SARS-CoV-2 RNA positivity from an oral or nasal swab, as measured by a nucleic acid amplification test, documented positive antigen testing, or positive nucleocapsid antibody. Documentation of the positive test is required.
3. Presence of persistent symptoms, defined as at least one COVID-attributed symptom newly present during acute illness or worse than baseline and reported to still be present for at least 90 days following symptom onset. This will be ascertained using study case report forms.
4. Reduced exercise capacity <100% predicted or self-reported reduction in exercise capacity compared to pre-COVID.
5. Willing and able to actively participate in cardiac rehabilitation including attending at least 12 in person sessions at UCSF Parnassus (intervention arm only).
6. Agree to participate in the LIINC Study including the cardiovascular substudy if they are not already participating.

Exclusion Criteria:

1. Pregnant or intention to become pregnant during study
2. Pre-existing congenital heart disease, heart failure, pulmonary hypertension, heart or lung transplant, or cardiac valve surgery
3. Myocardial infarction, or coronary artery bypass graft surgery, or new diagnosis of heart failure with a reduced ejection fraction <40% within 90 days prior to enrollment (Class I indications for cardiac rehabilitation)
4. Acute myocarditis diagnosed <90 days prior
5. Atrial fibrillation, atrial flutter, or other arrhythmias requiring antiarrhythmic therapy
6. Use of beta-blockers, non-dihydropyridine calcium channel blockers or ivabradine
7. Implanted pacemaker or defibrillator
8. Chronic lung disease requiring the use of home oxygen therapy
9. Inability to ride a sitting bicycle for CPET
10. Severe post-exertional malaise or symptom worsening that would preclude participation in cardiac rehabilitation
11. Medical or psychological comorbidities that would prevent safe participation in the trial, in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in adjusted heart rate reserve | Baseline and 12 weeks
  Adjusted heart rate reserve (peak HR-rest HR)/(220-age-rest HR) achieved during symptom-limited maximal cardiopulmonary testing performed with cycle ergometer
Change in Peak VO2 (ml/kg/min) | Baseline and 12 weeks
  Peak VO2 measured with maximal symptom limited cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Change in Peak VO2 (percent predicted) | Baseline and 12 weeks
  Peak VO2 (percent predicted using the Wasserman equations) measured with maximal symptom limited cardiopulmonary exercise testing
Number of Cardiac Rehabilitation sessions attended | 12 weeks
  Number of in person and virtual sessions attended by each participant
Change in Proportion with peak VO2 less than 85% predicted | Baseline and 12 weeks
  Proportion with peak VO2<85% predicted (using the Wasserman equations) measured with maximal symptom limited cardiopulmonary exercise testing
Change in Number of Long COVID symptoms | Baseline and 12 weeks
  Long COVID symptoms assessed using the LIINC symptom questionnaire (number of symptoms, more symptoms is worse).
Change in Composite Autonomic Symptom Scale-31 (Compass 31) Score | Baseline and 12 weeks
  Compass 31 summary score (0-100, with higher score indicating more severe autonomic symptoms).
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline and 12 weeks
  The PHQ-9 is a self-administered diagnostic instrument for depression. The PHQ-9 score ranges from 0 to 21, with higher scores indicating more severe depression.
Change in Generalized Anxiety Disorder Screener (GAD-7) Score | Baseline and 12 weeks
  The GAD-7 is a self-administered diagnostic instrument for depression. The GAD-7 score ranges from 0 to 27, with higher scores indicating more severe anxiety.
Change in Short Form Survey (SF-36) Score | Baseline and 12 weeks
  Overall quality of life using the short form health survey (SF-36). Scores range from 0-100 with higher scores representing a more favorable health state. The 36 questions are combined to form 8 scales in the domains of physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
Change in Quality of life assessed with EuroQol (EQ-5D) Visual Analogue Scale | Baseline and 12 weeks
  Quality of life on EQ-5D VAS (0-100, with 100 being the best).
Change in Inflammation | Baseline and 12 weeks
  hsCRP (mg/L) is a marker of inflammation
Net Promotor Score | 12 weeks
  Would you recommend cardiac rehabilitation to your family/friends (1-10 scale). The percentage who report 0-6 ("detractors") is subtracted from the percentage who report 9 or 10 ("promotors") to calculate a "Net Promoter Score."

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Durstenfeld, MD MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No